CLINICAL TRIAL: NCT04753645
Title: The Effect of Public Handwashing Stations on Health Behaviour and Outcomes During COVID-19
Brief Title: BRAC Institute of Governance and Development-Hygiene Behavioural Change and Coalition
Acronym: (BIGD-HBCC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BRAC University (Other)
Collaborators: The Behavioural Insights Team (Other); Brac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: BIGD2021
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hygiene Practices and Knowledge
Keywords: Handwashing station; mask usage; behvaioural change
MeSH Terms: interventions — Soaps

STUDY DESIGN:
Intervention Model Description: From each of 20 sub-district, out of potential villages for a public handwashing stations (HWS) we randomly selected 10 villages, of which 5 are assigned to control group or non-HBCC intervention villages and 5 are assigned to treatment group receiving the interventions. We have 98 control and 96 treatment villages due to an insufficient number of selected villages in one sub-district. First round survey revealed significant increase in soap use and not-significant decrease in handwashing (HW) frequency and soap expenditure. Our hypothesis is that there might be causality between HW and soap use. To test this, we provide soap to randomly selected 50% of our surveyed households, stratified at the sub-district level. 1,909 and 1,933 hhs from treatment and control villages received soap. Due to nationwide lockdown, we conducted follow-up phone survey. Also, to minimize Ramadan effect, we randomly divided the sample into two groups- to be surveyed before (44%) and during Ramadan (56%).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HBCC and no soap (Experimental): BRAC has built 1000 handwashing stations in 20 sub-districts from 3 divisions (out of a total of 8 divisions), namely Dhaka, Mymensingh and Khulna, to increase the access of communities to handwashing facilities. In addition to these handwashing stations, there are other supports available in the intervention areas i.e. in-person demonstration, hygiene meetings, and soap distribution from BRAC. However, this group did not receive any soap from the research team.
  Interventions: Behavioral: Handwashing stations at the public places and no soap
- No HBCC project and no soap (Experimental): In these randomly selected villages, BRAC did not implement any activity of its HBCC project. Also, the research team did not distribute soap to these households
  Interventions: Behavioral: No activities of the HBCC project and also no soap (Pure Control)
- Soap received but no HBCC (Experimental): In these randomly selected villages, BRAC did not implement any activity of its HBCC project but the research team randomly selected this group for soap distribution.
  Interventions: Behavioral: Soap distributed but no activities of the HBCC project
- Both HBCC project and Soap received (Experimental): These households belong to those villages where the HBCC project has been implemented and also received the soap from the research team.
  Interventions: Behavioral: HBCC project and Soap

INTERVENTIONS:
Behavioral: Handwashing stations at the public places and no soap — BRAC has built 1000 handwashing stations in 20 sub-districts from 3 divisions (out of a total of 8 divisions), namely Dhaka, Mymensingh and Khulna, to increase the access of communities to handwashing facilities. In addition to these handwashing stations, there are other supports available in the intervention areas i.e. in-person demonstration, hygiene meetings, and soap distribution from BRAC. However, this group did not receive any soap from the research team.
  Other Names: In-person demonstration
  Arms: HBCC and no soap
Behavioral: No activities of the HBCC project and also no soap (Pure Control) — In these randomly selected villages, BRAC did not implement any activity of its HBCC project. Also, the research team did not distribute soap to these households
  Arms: No HBCC project and no soap
Behavioral: Soap distributed but no activities of the HBCC project — In these randomly selected villages, BRAC did not implement any activity of its HBCC project but the research team randomly selected this group for soap distribution.
  Arms: Soap received but no HBCC
Behavioral: HBCC project and Soap — These households belong to those villages where the HBCC project has been implemented and also received the soap from the research team.
  Arms: Both HBCC project and Soap received

SUMMARY:
In line with BRAC's overall goals to limit the COVID19 transmission, BRAC has constructed 1,000 handwashing stations coupled with other supports i.e. in-person demonstration, hygiene meetings, and soap distribution in Bangladesh. The purpose of this study is to assess the impact of public handwashing stations (HWSs) on people's hygiene behavior and health outcomes in response to the COVID-19 situation. For this, at the household level, we will collect information on self-reported handwashing practices, income, health status, and HWSs along with other relevant socio-demographic variables in detail. In addition, we will observe people's mobility, mask usage at public places, and the HWSs usage; and will associate the observed HWSs usage with their self-reported health outcomes. This study will conduct surveys on households (7,760) and public (5,820) in 20 sub-districts of Mymensingh, Khulna, and Dhaka divisions.

Overall, this study is expected to directly benefit study participants and their communities by unveiling new evidence to inform BRAC's existing hygiene behavioral change programming in these communities. In addition, this information will yield future societal benefits by generating evidence on how to effectively implement and disseminate infrastructure and information that people can trust, believe, and use to form healthy hygiene habits.

DETAILED DESCRIPTION:
In line with the overall goals of HBCC for reducing the transmission of COVID-19 via rapid response interventions to raise awareness and enacting long-term behaviour change regarding people's personal and environmental hygiene habits, BRAC has taken an adaptive approach under the Hygiene and Behaviour Change Collation (HBCC) platform. The aim of this project is to systematically change the behaviour of people across communities in Bangladesh via interventions such as setting up handwashing stations and broadcasting behaviourally-informed messages to nudge people to adopt healthier prevention and response practices.

To achieve the overall goals of the project and positively impact the lives of over 10 million people in communities across Bangladesh, BRAC primarily chose 20 sub-districts from 3 divisions (out of a total of 8 divisions) for implementing the interventions, namely Dhaka, Mymensingh and Khulna. The prime activity is to install 1,000 handwashing stations across these sub-districts to increase the access of communities to handwashing facilities. The BRAC handwashing stations have been designed to enhance both availability and inclusiveness, fitted with foot-operated pedals for dispensing water and liquid soap, to reduce contact with sink surfaces and thereby reduce probability of transmission from the device surface. They have been fitted with posters, promoting handwashing with proper technique, and have also been designed to allow hand-washers to maintain social distance while using the devices.

In addition to these handwashing stations, there are other supports available in the intervention areas i.e. in-person demonstration, hygiene meetings, and soap distribution. After the economy opened up in Bangladesh after a long lockdown, the community engagement activities in the form of in-person communication and forum discussions, to motivate people to uptake safe hygiene behaviours including but not limited to regular handwashing. In these demonstrations and meetings, the participants are motivated to adopt recommended hygiene behaviours such as handwashing with soap, mask usage and disposal, sneezing etiquette, social distancing, etc. Along with the BRAC staff, the WASH entrepreneurs who are members of the local community whom BRAC traditionally supports with free training in entrepreneurship and market development to improve the communities' access and knowledge of hygiene products. The HBCC project empowers them with responsibilities to disseminate the messages of the recommended behaviours and distribute the soap in the communities across the intervention areas, especially the poorest of the poor community and the participants who attend the meetings regularly.

Primary Outcomes (end points)

The main outcome variables of interest in this study are:

i) daily handwashing frequency ii) likelihood of using soap when handwashing iii) prevalence of transmissible diseases in the past 15 days Primary Outcomes (explanation) i) constructed using the self-reported daily frequency of handwashing and typical handwashing times ii) constructed using self-report (times out of 10), rapid observation of the presence of soap near handwashing facilities, and self-reported expenditure on soap iii) constructed using self-report of symptoms and specific diseases Secondary Outcomes i) knowledge of handwashing practices ii) attitudes towards handwashing iii) use of public handwashing stations and alternatives to public handwashing stations iii) frequency of mask-wearing

ELIGIBILITY:
Inclusion Criteria:

* Must live in the villages where BRAC is implementing the interventions

Exclusion Criteria:

-

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3840 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Daily handwashing frequency | One day
  Constructed using the self-reported daily frequency of handwashing and typical handwashing times
Likelihood of using soap when handwashing | One day
  Constructed using self-report (times out of 10), rapid observation of the presence of soap near handwashing facilities, and self-reported expenditure on soap
Prevalence of transmissible diseases in the past 15 days | In last 15 days
  Constructed using self-report of symptoms and specific diseases

SECONDARY OUTCOMES:
Knowledge of handwashing practices | 3 months
  Self-reported knowledge on handwashing practices
Attitudes | 3 months
  Attitudes towards handwashing
Handwashing at the public places | 3 months
  Use of public handwashing stations and alternatives to public handwashing stations
Mask usage | 3 months
  Frequency of mask-wearing

CONTACTS AND LOCATIONS:
Locations (1):
- BRAC, Bangladesh, Dhaka, Bangladesh